CLINICAL TRIAL: NCT03297242
Title: A Retrospective Study of the Efficacy of Compound Lactobacillus Acidophilus Combined With Bismuth Quadruple Rescue Therapy on Patients With H Pylori Eradication Failures
Brief Title: Study the Effect of Probiotics Combined With Bismuth Quadruple Rescue Therapy on H Pylori Infective Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, director of the Digestive Department, Changhai Hospital
Other Study IDs: chbs230023
Record Dates: First submitted 2017-09-23; First posted 2017-09-29 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori eradication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospectivly follow-up the outpatients for H pylori eradication failures more than 2 times in the digestive department of Changhai hospital from 2015-2017,analyse the eradication rates and adverse effects of the therapy with 2w's compound lactobacillus acidophilus followed by 10d's bismuth, furazolidone, tetracycline contained quadruple scheme.

DETAILED DESCRIPTION:
H pylori infection rate has been up to half of the world population. H pylori infection is associated with various diseases, especially gastric cancer.

With the increasingly resistant to antibiotics,the eradication rate has decreased a lot with traditional triple therapy. Exploring a valid scheem for patients who have failed multiple times is important.

Probiotics can improve gastrointestinal microenvironment, then release the adverse effects during the eradication process.Additionally,there is also a lot evidence that probiotics can inhibit H plori，but still controversially.

There is a low resistant rate about furazolidone and tetracycline. In this study investigators observe the efficacy of the therapy 2w's compound lactobacillus acidophilus followed by 10d's bismuth, furazolidone, tetracycline contained quadruple scheme on patients who have failed more than 2 times. 4 to 6 weeks after the therapy, if Urea Breath Test (UBT) is nedative which means eradicating H plori successfully.

ELIGIBILITY:
Inclusion Criteria:

* H pylori eradication had failed more than 2 times
* Patients had never used furazolone and tetracycline
* The age varied from 18 to 80 years old

Exclusion Criteria:

* H pylori initial eradication or had failed only 1 time
* The age was lower than 18,or higher than 80 years old
* Patients who had serious heart pulmonary disease ,live renal disease, or any cancers
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mainland in China
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
urea breath test | 4-6 weeks after the quadruple therapy
  if urea breath test is negative,it means H pylori eradicated successfully

SECONDARY OUTCOMES:
adverse effects | 1month
  adverse effects mean the new symptoms during the treatment process,such as nausea,vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao S Li, MD, Principal Investigator